CLINICAL TRIAL: NCT03559725
Title: Evaluation of the Abuse Liability of Very Low Nicotine (VLN) Mentholated Cigarettes With Characterization of Nicotine Exposure Profiles in Adult Smokers
Brief Title: Evaluation of Abuse Liability of Very Low Nicotine (VLN) Mentholated Cigarettes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 22nd Century Group, Inc. (Industry)
Collaborators: Vince & Associates Clinical Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CEG-P1-078
Record Dates: First submitted 2018-05-23; First posted 2018-06-18 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Tobacco Use
Keywords: Abuse liability
MeSH Terms: conditions — Tobacco Use | interventions — Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: In part A each subject will have the opportunity to use either their own brand cigarette, nicotine gum or VLN menthol cigarettes ad libitum for 4 hours after which they will answer a questionnaire on using the product again. In Part B the subjects will have a controlled use session with each product followed by and uncontrolled session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VLN Menthol Cigarettes (A) (Experimental): Subjects will smoke VLN menthol cigarettes
  Interventions: Other: Usual Brand Menthol Cigarettes (B); Drug: Nicotine gum (C)
- Usual Brand Menthol Cigarettes (B) (Experimental): Subjects will smoke their usual brand menthol cigarettes
  Interventions: Other: VLN menthol cigarettes (A); Drug: Nicotine gum (C)
- Nicotine Gum (C) (Experimental): Subjects will chew nicotine gum
  Interventions: Other: VLN menthol cigarettes (A); Other: Usual Brand Menthol Cigarettes (B)

INTERVENTIONS:
Other: VLN menthol cigarettes (A) — 0.4mg nicotine / g tobacco king size filter menthol cigarette
  Arms: Nicotine Gum (C); Usual Brand Menthol Cigarettes (B)
Other: Usual Brand Menthol Cigarettes (B) — Usual brand king size menthol cigarettes
  Arms: Nicotine Gum (C); VLN Menthol Cigarettes (A)
Drug: Nicotine gum (C) — 4 mg nicotine gum
  Arms: Usual Brand Menthol Cigarettes (B); VLN Menthol Cigarettes (A)

SUMMARY:
This study is designed to evaluate the abuse liability of mentholated very low nicotine cigarettes compared to nicotine gum and usual brand cigarettes.

DETAILED DESCRIPTION:
This study will be a randomized, two-part, 3-way crossover designed to evaluate the abuse liability, pharmacokinetics (PK), and product use behavior associated with study products, including menthol VLN cigarettes, subjects' own-brand cigarettes, and nicotine polacrilex gum in healthy adult male and female exclusive smokers. Subjects will participate in a standard Screening visit and one 7-day Confined Assessment Phase, which will include a product trial session (Day -1), and two study parts (Part A and Part B). Following the Screening visit, eligible subjects will check-in to the study site on Day -1. Following the polacrilex gum training session, subjects will be required to abstain from nicotine- and tobacco-containing products for approximately 20 hours until the first product use session on Days 1 to 3; use of other nicotine-containing products will be prohibited throughout the study. No additional tobacco or nicotine products will be provided after the second product use on Days 4 to 6.

On Day 1, subjects will be randomized to one of three product sequence groups in Part A, which will consist of an ad libitum product use session for each of the following study products for 4 hours in a randomized crossover manner (Days 1 to 3; one product per day):

Product A: VLN menthol cigarette

Product B: Own-brand filtered standard king size menthol cigarette

Product C: 4 mg Nicotine polacrilex gum

A pharmacodynamic measure ("use product again" visual analog scale (VAS)) will be administered at the end of each ad libitum product use period. Product use behaviors (i.e., number of units consumed,duration of gum in mouth) will be collected throughout each ad libitum product use period. Upon completion of Part A, subjects will be randomized to one of three product sequence groups in Part B, which will consist of 3 study days (Days 4 to 6), with one product per day. Each study day will consist of: 1) Controlled Product Use Session (10 puffs from their own-brand cigarette or VLN menthol cigarette [maximum 3 ± 2 seconds per puff] at approximately 30 ± 5-second interpuff intervals, or chew the nicotine polacrilex gum using the "chew and park" method for 10 minutes); and 2) Uncontrolled Product Use Session (ad libitum use for 10 minutes). The Controlled Product Use Session and Uncontrolled Product Use Session will be separated by approximately 6 hours. During Part B, pharmacodynamic measures, pharmacokinetics (PK) , and product use behavior (Uncontrolled only) will be collected at various time points each day.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be required to meet each one of the following inclusion criteria in order to be eligible for participation in the study:

1. Must provide written informed consent prior to the initiation of any protocol-specific procedures.
2. Male and female adults, between 22 to 65 years of age, inclusive.
3. Body mass index (BMI) within 18.0 to 35.0 kg/m2, inclusive (minimum weight of at least 50.0 kg at Screening).
4. Healthy, as determined by no clinically significant medical history, physical examination, 12-lead ECG, vital signs or laboratory (including hematology, clinical chemistry, urinalysis, and serology) findings at Screening, as judged by an investigator.
5. Smoking history of an average of at least 10 manufactured filtered standard (i.e., not slim) king size combustible cigarettes daily for at least 1 year prior to Screening. Brief periods (i.e., up to 7 consecutive days) of non-smoking during the 3 months prior to Screening (e.g., due to illness or participation in a study where smoking was prohibited) will be permitted.
6. Self-reporting of desire to smoke within approximately 30 minutes of waking.
7. Positive urine cotinine (≥500 ng/mL) at Screening.
8. Negative pregnancy test at Screening and Day -1 (check-in) for all female subjects.
9. Female subjects of non-childbearing potential must be surgically sterile or 1 year postmenopausal (as confirmed by serum Follicle Stimulating Hormone (FSH) > 35 U/L). A subject is considered to be surgically sterile if she has had a tubal ligation, hysterectomy, bilateral salpingo-oophorectomy or bilateral oophorectomy, or hysterectomy with bilateral salpingo-oophorectomy. If the subject is of childbearing potential, she must be using a medically accepted method of contraception and agree to continued use of this method for the duration of the study and for 30 days after completion of the study. Acceptable methods of contraception include abstinence, birth control pill, or an intrauterine device (known to have a failure rate of less than 1% per year) or double barrier method of contraception (e.g., male condom in addition to a diaphragm, contraceptive sponge or spermicide).
10. Able to speak, read, and understand English sufficiently to allow completion of all study assessments.
11. Must be willing to comply with the requirements and restrictions of the study.

Exclusion Criteria:

Subjects will not be eligible to participate in this study if any one of the following exclusion criteria is met:

1. Inability to tolerate 4 mg nicotine polacrilex gum during product use trial on Day -1 (check-in) or dentition prevents subjects from chewing gum.
2. History or presence of any clinically significant cardiac, psychiatric, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal, or other major disease at Screening, which in the opinion of an investigator would jeopardize the safety of the subject or the validity of the study results.
3. History or presence of any type of malignant tumors.
4. Clinically significant abnormal findings on the vital signs, physical examination (including oral exam), medical history, or clinical laboratory results, in the opinion of an investigator.
5. Positive serology test results for human immunodeficiency virus (HIV-1/HIV-2) Antibodies, hepatitis B surface antigen (HbsAg), or hepatitis C Antibody (HCVAb).
6. An acute illness (e.g., upper respiratory infection, viral infection) requiring treatment within 2 weeks prior to Day -1 (check-in).
7. Drug or alcohol abuse or dependence within the 24 months prior to Screening (except nicotine), as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition text revision (DSM-IV-TR), or any self-reported dependence or "addiction" within the subject's lifetime (except nicotine or caffeine).
8. Subjects who have ever been in treatment for substance use disorder(s) or who are currently
9. Positive urine drug screen (UDS) or urine alcohol test at Screening or Day -1 (check-in).
10. History or any current conditions that may interfere with drug absorption, distribution, metabolism, or excretion.
11. History of severe allergic reaction (including anaphylaxis) to any substance, or previous status asthmaticus, or food allergies/intolerances/restrictions, or special dietary needs which, in the judgment of an investigator, contraindicates the subject's participation in the study.
12. Requires concomitant treatment with prescription or non-prescription products that contain pseudoephedrine (e.g., nasal/sinus decongestants).
13. Self-reported use of nicotine polacrilex gum, or other nicotine replacement therapy products in the 30 days prior to Day -1 (check-in). Isolated incidents within 30 days prior to Day -1 (check-in) may be permitted at the discretion of the investigator.
14. Subject has unsuitable or difficult venous access or is unwilling or unable to undergo direct venipuncture or catheter insertion.
15. Subject has donated or lost 100 to 499 mL whole blood within 30 days or more than 499 mL whole blood within 56 days preceding entry into the Confined Assessment Phase.
16. Subject is an employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member defined as a spouse, parent, child or sibling, whether biological or legally adopted.
17. Subject is lactating and or breast feeding.
18. A subject who, in the opinion of an investigator, is considered unsuitable or unlikely to comply with the study protocol for any reason.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Emax_urge(controlled) | 3 days - administered at the end of each product use session (Use of each product on a different day)
  The maximum reduction in Visual Analog Scale (VAS) score for the question "Urges to smoke" (Tobacco/Nicotine Withdrawal Questionnaire) between pre-use and post-use (i.e., VASpre-use1 - VASpost-use1) during the first product use in Part B.

SECONDARY OUTCOMES:
Cmax(controlled); Maximum Nicotine Concentration | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Maximum measured plasma nicotine concentration during the Controlled Use Session.
T1/2(controlled); Terminal Half Life | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Apparent first-order terminal nicotine elimination half-life calculated as 0.693/Kel of the plasma concentration-time curve from time zero (defined as the start of controlled use) to 180 minutes
Kel(controlled); Elimination Rate Constant | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Apparent first-order terminal nicotine elimination rate constant calculated from a semi-log plot of the plasma concentration-time curve of the Controlled Use Session.
Tmax(controlled); Maximum Time | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Time of the maximum measured plasma nicotine concentration during the Controlled Use Session.
AUC(controlled); Area under the nicotine concentration-time curve | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Area under the nicotine concentration-time curve calculated using linear trapezoidal summation from time zero (defined as the start of controlled use) to 180 minutes (or the last quantifiable concentration during that interval).
Cmax(uncontrolled); Maximum Nicotine Concentration | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Maximum measured plasma nicotine concentration during the Uncontrolled Use Session.
T1/2(uncontrolled); Terminal Half Life | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Apparent first-order terminal nicotine elimination half-life calculated as 0.693/Kel of the plasma concentration-time curve from time zero (defined as the start of uncontrolled use) to 540 minutes.
Kel(uncontrolled); Elimination Rate Constant | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Apparent first-order terminal nicotine elimination rate constant calculated from a semi-log plot of the plasma concentration-time curve of the Controlled Use Session.
Tmax(uncontrolled); Maximum Time | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Time of the maximum measured plasma nicotine concentration during the Uncontrolled Use Session.
AUC(uncontrolled); Area under the nicotine concentration-time curve | Pre, 2,5,7,10,12,15,20,30,45,60,90,120,150, and 180 minutes
  Area under the nicotine concentration-time curve calculated using linear trapezoidal summation from time 360 (defined as the start of uncontrolled use) to 540 minutes (or the last quantifiable concentration during that interval).
Emax_urge (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minute
  The largest VAS score recorded for the response to "Urges to Smoke" (Tobacco/nicotine withdrawal questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_anx (Controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Urges to Smoke" (Tobacco/nicotine withdrawal questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_anx (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Anxious" (Tobacco/nicotine withdrawal questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_diffct (Controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Difficulty Concentrating" (Tobacco/nicotine withdrawal questionnaire) during the product use in Controlled Section of Part B.
Emax_diffct (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Difficulty Concentrating" (Tobacco/nicotine withdrawal questionnaire) during the product use in Controlled Section of Part B.
Emax_impat (Controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Impatient" (Tobacco/nicotine withdrawal questionnaire) during the product use in Controlled Section of Part B.
Emax_impat (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Impatient" (Tobacco/nicotine withdrawal questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_crav (Controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Craving a Cigarette" (Tobacco/nicotine withdrawal questionnaire) during the product use in Controlled Section of Part B.
Emax_crav (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Craving a Cigarette" (Tobacco/nicotine withdrawal questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_plas (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Pleasant" (Direct effects of product questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_stf (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Satisfying" (Direct effects of product questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_stf (Controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Satisfying" (Direct effects of product questionnaire) during the product use in Controlled Section of Part B.
Emax_calm (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Calm" (Direct effects of product questionnaire) during the product use in Controlled Section of Part B.
Emax_calm (Controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Calm" (Direct effects of product questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_conc (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Concentrate" (Direct effects of product questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_conc (controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Concentrate" (Direct effects of product questionnaire) during the product use in controlled Section of Part B.
Emax_awake (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Awake" (Direct effects of product questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_awake (controlled) | pre, 5, 15, 30, 60, and 90 minutes
  he largest VAS score recorded for the response to "Awake" (Direct effects of product questionnaire) during the product use in controlled Section of Part B.
Emax_sick (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Sick" (Direct effects of product questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_sick (Controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Sick" (Direct effects of product questionnaire) during the product use in Controlled Section of Part B.
Emax_hunger (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Hunger" (Direct effects of product questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_hunger (Controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "Hunger" (Direct effects of product questionnaire) during the product use in Controlled Section of Part B.
Emax_more (Uncontrolled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "More" (Direct effects of product questionnaire) during the product use in Uncontrolled Section of Part B.
Emax_more (Controlled) | pre, 5, 15, 30, 60, and 90 minutes
  The largest VAS score recorded for the response to "More" (Direct effects of product questionnaire) during the product use in Controlled Section of Part B.
Inhalations | 3 product use days (Use of each product on a different day)
  Number of product inhalations (cigarettes only) during uncontrolled use sessions
Puff durations | 2 product use days (Use of each product on a different day)
  Duration of inhalations (cigarettes only) during uncontrolled use sessions
Gum durations | 1 product use day
  Duration of gum in mouth during uncontrolled use sessions
Use Product Again | 1 product use day
  The VAS score recorded for the response to "Use Product Again" (Use product again questionnaire) during the ad libitum product use in Part A.
Emax_plst(controlled) | 3 days - administered at the end of each product use session (Use of each product on a different day)
  The largest VAS score recorded for the response to the question "Is the product "Pleasant" right now?" (Direct Effects of Product Questionnaire) during the first product use in Part B

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Vince and Associates Clinical Research, INC
Locations (1):
- Vince and Associates Clinical Research, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT03559725/Prot_000.pdf